CLINICAL TRIAL: NCT04232917
Title: Randomized, Placebo-controlled, Double-blind Study to Evaluate 2LPAPI® Efficacy on the Clearance of Genital HR-HPV Infections.
Brief Title: Study of 2LPAPI® on the Clearance of Genital HR-HPV Infections.
Acronym: PAPION
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Labo'Life (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LLB-2017-01
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Human Papilloma Virus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2LPAPI® arm (Experimental): The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment. The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Interventions: Drug: 2LPAPI®
- Placebo arm (Placebo Comparator): The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment. The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2LPAPI® — Treatment
  Other Names: 2LPAPI
  Arms: 2LPAPI® arm
Drug: Placebo — Placebo
  Arms: Placebo arm

SUMMARY:
Human papillomavirus (HPV) is a prevalent pathogen, the epidemiology of which has mostly been studied in the uterine cervix and the vagina.

The KCE Report 238Cs (2015) recommends " HR-HPV-positive women should not be offered colposcopy immediately. Triage should be done using cytology for this purpose. If cytological abnormalities (ASCUS+) are found, immediate referral should follow for diagnosis and, where appropriate, treatment. If no abnormalities are observed in triage, the subject should be offered follow-up testing (cytology) at six months. ".

There is no treatment that is recommended during this lap time. The 2LPAPI® has been available for more than 20 years, and has received a marketing authorization in Belgium by the FAMHP. It is used as an immune regulator in the treatment of HR-HPV infections. Since 2LPAPI® has been made available, clinical observational data collected on treated patients have shown the beneficial effect on the clearance of HPV.

The purpose of this placebo-controlled trial is to evaluate the efficacy of 2LPAPI® on the clearance of genital HR-HPV infections.

DETAILED DESCRIPTION:
The study duration will be 72 months with 60 months of inclusion (that may be extended if the expected number of patients is not reached after 60 months) and 12 months of follow-up.

Patients aged between 25 and 45 years presenting a diagnosis of HR-HPV infection during the routine screening visit for cervical cancer prevention.

The total number of patients to include will be 284 with 142 patients per group.

Primary objective:

Comparison of the efficacy of 2LPAPI® versus placebo on the clearance of genital HR-HPV infections after 12 months of follow-up.

Secondary objectives:

Comparison of 2LPAPI® versus placebo on:

* HR-HPV infection clearance rate at 6-month visits,
* HR-HPV infection clearance rate by HPV type at 6-month and 12-month visits,
* Evolution of cytology,
* Normalization of cytology for the subpopulation of patients with a baseline non normal cytology,
* Safety: adverse events (AEs) and serious adverse events (SAEs), considered as related or not to the study drug.

Treatment phase:

Group n°1 = 2LPAPI® (6 months of treatment) Group n°2 = Placebo (6 months of treatment) Post-treatment follow-up phase: 6 months. Treatment will be considered successful if the clearance of HR-HPV is done and the cytology is normal.

ELIGIBILITY:
Inclusion Criteria:

* Women 25-45 years,
* Women of childbearing age under effective contraception,
* Patient with last cytology less than 3 years and normal or not more than LSIL or CIN I at the histology,
* Patient with current cytology presenting normal, ASC-US, AGUS, LSIL, ASC-H, AGC or LSIL+ASC-H results or current diagnosis of CIN I at the histology,
* Patient with HR-HPV diagnosis at the current cervical collection,
* Patient reporting a current stable sexual relationship (steady sexual partner during study duration),
* Patient having faculties to understand and respect the constraints of the study,
* Signature of the Informed Consent Form.

Exclusion Criteria:

* Pregnant or breastfeeding woman,
* Patient presenting HSIL diagnosis at the cytology or CIN II or CIN III diagnosis at the histology,
* Patient having received HPV vaccination in the last month,
* Patient previously subject to total hysterectomy,
* Patient under immunotherapy (including immunosuppressive treatment) or micro-immunotherapy received during last previous 6 months,
* Patient with known lactose intolerance,
* Patient who participated in a clinical study in the previous 3-months' period,
* Patient who is not sufficiently motivated to engage in a follow-up period of 12 months, or likely to travel or to move before the end of the study,
* Patient with severe immunodeficiency disease requiring long term treatment (*) or under chemotherapy or radiotherapy,
* Patient under listed homeopathic or phytotherapy treatment (see protocol),
* Patient using or addicted to recreational drugs.

(*) important renal or respiratory insufficiency, transplanted or grafted patients, HIV/AIDS, terminal cancer.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 284 (Estimated)
Dates: Start 2020-10-17 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the efficacy of 2LPAPI® versus placebo on the clearance of genital HR-HPV infections after 12 months of follow-up. | 12 months
  The primary objective of the study will be to compare the number of patients with positive HR-HPV infection status observed at 12 months and the number of patients with positive HR-HPV infection status observed at the inclusion.

SECONDARY OUTCOMES:
Comparison of 2LPAPI® versus placebo on HR-HPV infection clearance rate at 6-month visits. | 6 months
  The objective of this outcome will be to compare the number of patients with positive HR-HPV infection status observed at 6 months and the number of patients with positive HR-HPV infection status observed at the inclusion.
Comparison of 2LPAPI® versus placebo on HR-HPV infection clearance rate by HPV type at 6-month and 12-month visits. | 6 and 12 months
  The objective of this outcome will be to compare the number of patients with specific type of HPV infection observed at 6 and 12 months and the number of patients with specific HPV infection status observed at the inclusion.
Evolution of cytology (normalization, stagnation or worsening) at 6-month and 12-month visits. | 6 and 12 months
  The objective of this outcome will be to compare the evolution of the cytology at 6-month and 12-month visits.
Normalization of cytology at 6-month and 12-month visits for the subpopulation of patients with a baseline non-normal cytology. | 6 and 12 months
  The objective of this outcome will be to compare the number of patients with a normal cytology at 6-month and 12-month visits in the subpopulation of patients with a baseline non-normal cytology.
Occurrence of adverse events (AEs) and severe adverse events (SAEs), considered as related or not to the study drug | 6 months

CONTACTS AND LOCATIONS:
Locations (11):
- Belgium (11):
  - CHU Saint-Pierre, Brussels
  - Clinique St Jean, Brussels
  - CHU Brugmann, Brussels
  - Hôpitaux Iris Sud - Iris Zuid Ziekenhuis, Brussels
  - Hôpital Civil Marie Curie ISPPC, Charleroi
  - Centre Hospital Reine Astrid Malmedy (CHRAM), Malmedy
  - Belgium, Namur
  - Cabinet privé, Namur
  - UCL Namur - site Sainte Elisabeth, Namur
  - Clinique Saint-Pierre Ottignies (CSPO), Ottignies
  - CHWAPI, Tournai